CLINICAL TRIAL: NCT06817915
Title: LMU Project on the Impact of Reviewing AI Annotated SD-OCT Therapy Assistance Reports on Ophthalmologists' Treatment Decision-making for Anti-VEGF Therapy in NAMD Patients
Brief Title: This Project At LMU Looks At How Using AI 2nd Opinion Report to Analyze Retinal Eye Scans Impact Doctors' Decisions About Treatment for Patients with a Specific Eye Disease (nAMD)
Acronym: LMU ASSIST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Schiefelbein (Other)
Collaborators: Deepeye Medical GmbH (Industry); Technomics Research (Industry); M3 Macula Monitor Muenster (Unknown)
Responsible Party: Sponsor-Investigator, Johannes Schiefelbein, Co-Project Lead, LMU Klinikum
Organization: LMU Klinikum (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2301LMUASSIST
Record Dates: First submitted 2025-01-27; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Neovascular Age-Related Macular Degeneration (nAMD)
Keywords: Decison-making; AI-Assisted treatment; artificial intelligence; clinical decision support; ophthalmology; SD-OCT; neovascular age-related macular degeneration; nAMD; anti-VEGF; explainable AI

STUDY DESIGN:
Intervention Model Description: Survey
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AI 2nd opinion assisted assessment of SD-OCT scan (Experimental): Ophthalmologists assess patient SD-OCT scans before and after reviewing AI-2nd opinion reports
  Interventions: Behavioral: AI assisted assessment of SD-OCT scans

INTERVENTIONS:
Behavioral: AI assisted assessment of SD-OCT scans — AI 2nd opinion report on nAMD treatment planning

SUMMARY:
This is a research plan from the University of Munich (LMU) that aims to study how the use of AI reports can impact ophthalmologists' decisions regarding treatment for patients with neovascular age-related macular degeneration (nAMD). This disease is a leading cause of vision loss, and while anti-VEGF treatments are effective, they require careful monitoring and retreatment decisions to maximize benefits.

The study will involve up to 1000 ophthalmologists with varying levels of expertise. These ophthalmologists will review SD-OCT scans and make treatment decisions before and after reviewing AI-generated reports. The primary objective is to compare these decisions and see how the AI reports influence them. Secondary objectives include assessing the accuracy and safety of the AI reports.

DETAILED DESCRIPTION:
This research project at LMU delves into the intersection of artificial augmentation and ophthalmology, specifically focusing on how AI-generated 2nd opinion reports can aid in the treatment planning of neovascular age-related macular degeneration (nAMD). The project will involve a diverse group of up to 1000 ophthalmologists, categorized into six user groups based on their expertise, ranging from residents to seasoned retina specialists.

The core of the research involves assessing the impact of AI-generated 2nd opinion reports on ophthalmologists' treatment decisions for nAMD. Participants will review SD-OCT scans and make initial treatment decisions. Subsequently, they will review AI-generated reports for the same scans and have the opportunity to revise their decisions. This process aims to evaluate the influence of AI insights on clinical judgment.

The project will be conducted virtually, with participants enrolling online from various countries. Data collection will be facilitated through an electronic system, ensuring efficiency and security. Statistical analysis will primarily involve descriptive statistics to summarize the findings. The results of the study will be disseminated through publication in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Electronically consented to the informed consent form (eICF)
* Criteria to be included in one of the following six Ophthalmology user groups:

Group 1 Non-retina specialist Group: Ophthalmology, completed ophthalmology residence with no or another subspecialty other than retina (e.g., Glaucoma, refractive, etc) Group 2 Resident Group: <5 years in residency in ophthalmology Group 3 Fellow Group: Retina specialist in training Group: in fellowship in vitreoretinal medicine, medical retina Group 4 Retina specialist Group: completed retina training, regular requalification Group 5 Junior reader Group: have already gained experience in the reporting clinical routine with the diagnostics in question and completed the initial certification process at an Image and Reading Center (acc. to centre's SOP) Group 6 Senior reader Group: specialist with several years of experience in the relevant field or have completed at least 3 years of residency training. Completed the certification process at the Image and Reading Center (acc. to centre's SOP)

Exclusion Criteria:

* Not an Ophthalmologist.
* Does not have time to participate in the estimated project duration of 30 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Ophthalmologist's Treatment Decision | There is only one survey filled out by the participant. In this survey, only one time point when participant views the SD-OCT and AI 2nd opinion report and fills out the survey questions.
  The number and percentage of initial treatment decisions that stayed the same after their review of the AI-CDS report The number and percentage of initial decisions that changed after their review of the AI-CDS report

SECONDARY OUTCOMES:
Performance Accuracy | There is only one survey filled out by the participant. In this survey, only one time point when participant views the SD-OCT and AI 2nd opinion report and fills out the survey questions.
  The number and percentage of correct assessments (accuracy) made by AI-CDS report vs image grading/reading center (M³ Macula Monitor Münster) assessment (control / gold standard / ground truth) The percentage of correct assessments (accuracy) made by each of the 6 user group vs. image grading and reading center (M³ Macula Monitor Münster) assessment (control / gold standard / ground truth).
  How often is the AI-CDS report correct? How often is each of the 6 user groups correct after viewing just the SD-OCT image?
  Intra-rater reliability:
  How often are ophthalmologists (each user group) right/wrong after viewing AI-CDS report and made any decision changes?
Safety prediciton assessment | There is only one survey filled out by the participant. In this survey, only one time point when participant views the SD-OCT and AI 2nd opinion report and fills out the survey questions.
  Yes/No prediction rates If an ophthalmologist is correct and AI-CDS report incorrect, how often does AI-CDS report mislead? Whether false-positive or false-negative? If an ophthalmologist is wrong and AI-CDS report correct, how often does AI-CDS report correct? Whether false-positive or false-negative?
Exploratory AI-CDS report Impact on Decision Making | There is only one survey filled out by the participant. In this survey, only one time point when participant views the SD-OCT and AI 2nd opinion report and fills out the survey questions.
  impact of AI-CDS report on ophthalmologist's decision-making survey

CONTACTS AND LOCATIONS:
Overall Officials: Director the Eye Clinic, Study Director — LMU Klinikum Eye Clinic
Locations (1):
- LMU Klinikum, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Chopra R, Preston GC, Keenan TDL, Mulholland P, Patel PJ, Balaskas K, Hamilton RD, Keane PA. Intravitreal injections: past trends and future projections within a UK tertiary hospital. Eye (Lond). 2022 Jul;36(7):1373-1378. doi: 10.1038/s41433-021-01646-3. Epub 2021 Jun 25. PMID 34172943